CLINICAL TRIAL: NCT02182934
Title: Efficacy of Ginsana in Improving Half-time Hemoglobin Re-oxygenation in Recreational Sports People: a Double-blind, Placebo Controlled Pilot Study
Brief Title: Efficacy of Ginsana in Improving Half-time Hemoglobin Re-oxygenation in Healthy Recreational Sports People
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1020.11
Record Dates: First submitted 2014-07-04; First posted 2014-07-08 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Healthy

ARMS (2):
- Ginsana (Experimental)
  Interventions: Drug: Ginsana
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ginsana
  Arms: Ginsana
Drug: Placebo
  Arms: Placebo

SUMMARY:
To assess the efficacy of Ginsana in improving hemoglobin re-oxygenation in healthy, recreational sports people and to assess the safety of the product.

ELIGIBILITY:
Inclusion Criteria:

* Male and female volunteers between 18 and 40 years old
* Females must test negative for pregnancy
* Recreational athletes according to the american college of sports medicine (ACSM) definition
* Familiar with the cycle ergometer exercise methodology
* Written inform consent according to good clinical practice (GCP) and local regulations

Exclusion Criteria:

* Pre treatment and/or concomitant treatment with any drug that any drug that may influence the trial symptomatology
* Alcohol and drug abuse as stated in the clinical trial manual
* Smokers
* Known hypertension
* Known hypercholesterolemia (moderate/severe)
* Female volunteers taking oral or injectable contraceptives
* Female volunteers of child bearing potential not using adequate means of birth control, other than contraceptive pills [intrauterine devices (IUDs)]
* Pregnancy and/or lactation
* Liver and/or renal and/or vascular disease
* Relevant allergy or known hypersensitivity to the investigational drug or its excipients
* Participation in another clinical trial within the last 4 weeks before the date of inclusion or concurrent participation in another clinical trial

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 1999-11; Primary Completion 2000-04 (Actual)

PRIMARY OUTCOMES:
Baseline-adjusted half-time hemoglobin re-oxygenation | day 84

SECONDARY OUTCOMES:
Baseline-adjusted half-time hemoglobin re-oxygenation | day 21, 42 and 63
maximum endurance time | day 21, day 42, day 63 and day 84
Change from baseline in respiratory threshold | Baseline, up to day 84
Change from baseline in thiobarbituric acid (TBARS) | Baseline, up to day 84
Change from baseline in glutathione superdismutase/glutathione superdismutase oxidised (GSG/GSSG) ratio | Baseline, up to day 84